CLINICAL TRIAL: NCT03907579
Title: Screen to Save: A Colorectal Cancer Educational Intervention
Acronym: S2S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Tracy L. Onega, Associate Director of Community Outreach and Education, Norris Cotton Cancer Center; Associate Professor, Dartmouth Geisel School of Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: D17190; P30CA023108-39 (NIH)
Record Dates: First submitted 2019-04-06; First posted 2019-04-09 (Actual); Results first posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Colorectal Cancer
Keywords: Knowledge
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inflatable colon educational module (Experimental): Participants attend a brief educational presentation in an inflatable colon, focused on colorectal cancer prevention and screening. Participants also receive a copy of the study information sheet and may receive written educational materials to take home. Participants complete a pre-test and a post-test to assess changes in knowledge and intention to get screened for colorectal cancer.
  Interventions: Behavioral: Inflatable colon educational module

INTERVENTIONS:
Behavioral: Inflatable colon educational module — Participants attend a brief educational presentation in an inflatable colon, learning about colorectal cancer prevention and screening.

SUMMARY:
The purpose of this research is to understand if an educational program about colorectal cancer helps improve people's knowledge of colorectal cancer prevention and screening and their intention to get screened for colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age: 50-74 years old
* Attendee at event where educational module is offered

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-03-11 (Actual); Primary Completion 2017-06-17 (Actual); Study Completion 2017-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Onega, PhD, MA, MS, Principal Investigator — Dartmouth College
Locations (1):
- Norris Cotton Cancer Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual de-identified data collected during the trial will be shared with the National Cancer Institute, Geographic Management of Cancer Health Disparities Program (GMaP) contacts, and NCI's designated contractor for the Screen to Save Initiative
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following data collection events
Access Criteria: For meta-analyses

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Inflatable Colon Educational Module
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Inflatable Colon Educational Module
Number analyzed (Participants) | 100
Age, Customized [Mean (Standard Deviation); unit: years] — Population: Two participants did not provide their age in the baseline survey.
  years
    Mean age: number analyzed (Participants) | 98
    Mean age | 59.5 (5.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 100
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 96
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 100
Correct Answers on Knowledge Questions [Mean (Standard Deviation); unit: correct answers] — Number of correct responses to a series of 14 true/false and multiple-choice test questions about colorectal cancer risks, prevention, and screening.
  correct answers | 10.78 (2.20)

OUTCOME MEASURES:

1. Primary Outcome: Change in Knowledge Related to Colorectal Cancer Risk, Prevention, and Screening
Description: A pre-test and post-test is conducted with participants to assess any changes in knowledge related to key learning outcomes expected from the educational intervention (assessed via 14 questions before and after learning).
Time Frame: Baseline and immediately following intervention
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Inflatable Colon Educational Module
Number analyzed (Participants) | 100
score on a scale | 1 [-4 to 6]
Statistical Analysis 1: Comparison: Inflatable Colon Educational Module; Test type: Superiority; p = 0.0001, Wilcoxon Signed Rank Test; z= -3.861

2. Primary Outcome: Number of Participants With Varying Levels of Behavioral Intentions Related to Colorectal Cancer Screening and Prevention
Description: Post-test conducted to assess behavioral intention related to five prevention and screening behaviors (assessed via 5 questions on a 4-point Likert scale, where a higher score indicates stronger behavioral intention). The scale for all behavioral intention measures started with, "As a result of the colorectal cancer screening information I received during the Screen to Save educational session, I am more likely to…"
Time Frame: Immediately following intervention
Population: Four intention questions were left blank/unanswered by one to two participants each.
Measure: Count of Participants; unit: Participants
Arm/Group | Inflatable Colon Educational Module
Number analyzed (Participants) | 100
Participants
  Intent to talk w/ provider about CRC screening: number analyzed (Participants) | 99
  Intent to talk w/ provider about CRC screening: Strongly agree | 71
  Intent to talk w/ provider about CRC screening: Agree | 28
  Intent to talk w/ provider about CRC screening: Disagree | 0
  Intent to talk w/ provider about CRC screening: Strongly Disagree | 0
  Intent to get screened for CRC: number analyzed (Participants) | 99
  Intent to get screened for CRC: Strongly agree | 67
  Intent to get screened for CRC: Agree | 30
  Intent to get screened for CRC: Disagree | 2
  Intent to get screened for CRC: Strongly Disagree | 0
  Intent to talk w/ family/friends about screening: number analyzed (Participants) | 98
  Intent to talk w/ family/friends about screening: Strongly agree | 64
  Intent to talk w/ family/friends about screening: Agree | 30
  Intent to talk w/ family/friends about screening: Disagree | 4
  Intent to talk w/ family/friends about screening: Strongly Disagree | 0
  Intent to eat healthier: number analyzed (Participants) | 99
  Intent to eat healthier: Strongly agree | 72
  Intent to eat healthier: Agree | 27
  Intent to eat healthier: Disagree | 0
  Intent to eat healthier: Strongly Disagree | 0
  Intent to increase physical activity: Strongly agree | 70
  Intent to increase physical activity: Agree | 29
  Intent to increase physical activity: Disagree | 1
  Intent to increase physical activity: Strongly Disagree | 0

ADVERSE EVENTS:
Time Frame: During presentation, up to 1 day
Arm/Group | Inflatable Colon Educational Module
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/79/NCT03907579/Prot_000.pdf
  • Informed Consent Form (2017-03-07): https://cdn.clinicaltrials.gov/large-docs/79/NCT03907579/ICF_001.pdf
  • Statistical Analysis Plan (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT03907579/SAP_002.pdf